CLINICAL TRIAL: NCT07407504
Title: An International, Multicenter, Open-label, Phase 1/2 Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics, and Efficacy of GenSci145, as Monotherapy or in Combination Therapy, in Participants With PIK3CA-mutated, Locally Advanced or Metastatic Solid Tumors.
Brief Title: GenSci145 as Monotherapy or in Combination Therapy, in Participants With PIK3CA-mutated, Locally Advanced or Metastatic Solid Tumors.
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GenSci145-101
Record Dates: First submitted 2026-02-03; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced or Metastatic Solid Tumors With PIK3CA-mutated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GenSci145 tablets (Experimental)
  Interventions: Drug: GenSci145 tablets

INTERVENTIONS:
Drug: GenSci145 tablets — Participants will receive GenSci145 as stipulated in the research protocol

SUMMARY:
An international, multicenter, open-label, Phase 1/2 clinical study to evaluate the safety, tolerability, pharmacokinetic characteristics, and efficacy of GenSci145, as monotherapy or in combination therapy, in participants with PIK3CA-mutated, locally advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
An international, multicenter, open-label, Phase 1/2 clinical study to evaluate the safety, tolerability, pharmacokinetic characteristics, and efficacy of GenSci145, as monotherapy or in combination therapy, in participants with PIK3CA-mutated, locally advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and voluntarily provide written ICF.
* Willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other protocol-specified procedures.
* Age 18-75 years (inclusive) at the time of providing informed consent.
* Disease diagnosis requirements:

Part 1:

1. Histologically or cytologically confirmed locally advanced or metastatic solid tumors.
2. Disease progression after standard therapy, or, in the opinion of the investigator, no available and effective standard therapy.

Part 2:

1. Histologically or cytologically confirmed HR+/HER2- locally advanced or metastatic breast cancer [HR+ is defined as estrogen receptor (ER) positive and/or progesterone receptor (PR) positive (≥10% of tumor cell nuclei showing positive staining); HER2- is defined as immunohistochemistry (IHC) 0 or 1+, or IHC 2+ with a negative in situ hybridization (ISH) result].
2. Disease progression after standard therapy, or, in the opinion of the investigator, no available and effective standard therapy.

Part 3 (doublet) and Part 4 Cohort 1:

1. Histologically or cytologically confirmed HR+/HER2- locally advanced or metastatic breast cancer.
2. Patients must meet one of the following:

   1. Disease progression during (neo)adjuvant endocrine therapy or within 12 months after completion of such therapy, without having received any prior therapy for metastatic disease.
   2. Disease progression occurring more than 12 months after completion of adjuvant endocrine therapy, followed by first-line endocrine therapy for metastatic disease, with subsequent progression on that therapy.
   3. Newly diagnosed advanced breast cancer with progression after first-line endocrine therapy.
3. Received ≤1 line of chemotherapy for advanced disease.
4. Prior use of CDK4/6 inhibitors must meet one of the following:

   1. Received CDK4/6 inhibitor therapy in the advanced setting with disease progression occurring during or within 12 months after treatment.
   2. Discontinued treatment due to intolerability caused by adverse reactions (e.g., hyperglycemia, rash).
   3. If not previously treated with a CDK4/6 inhibitor, a reasonable explanation must be provided (e.g., lack of drug availability).

Part 3 (triplet) and Part 4 Cohort 3:

1. Histologically or cytologically confirmed HR+/HER2- locally advanced or metastatic breast cancer.
2. Disease progression during adjuvant endocrine therapy with an aromatase inhibitor or tamoxifen, or within 12 months after completion of adjuvant endocrine therapy. If a CDK4/6 inhibitor was included as part of the (neo)adjuvant therapy, disease progression must occur >12 months after completion of CDK4/6 inhibitor therapy.

Part 4 Cohort 2:

1. Histologically or cytologically confirmed HR+/HER2- locally advanced or metastatic breast cancer with brain metastases; diagnosis and treatment requirements are consistent with those for Part 3 (doublet) and Part 4 Cohort 1.
2. No immediate need for CNS-specific treatment (e.g., radiotherapy or surgery), as determined by the investigator.

Part 4 Cohort 4:

1)Histologically or cytologically confirmed advanced solid tumors other than breast cancer, including but not limited to head and neck squamous cell carcinoma, gynecologic malignancies, or colorectal cancer.

2)Disease progression after standard therapy, or, in the opinion of the investigator, no available and effective standard therapy.

* Female participants enrolled in the breast cancer cohorts must meet one of the following conditions:

  1. Postmenopausal status, defined as any of the following:

     1. Surgical bilateral oophorectomy performed ≥14 days prior, with recovery to baseline status.
     2. Age ≥60 years.
     3. Age <60 years, amenorrhea ≥12 months, and follicle-stimulating hormone (FSH) and estradiol (E2) levels within the postmenopausal range according to local reference values, without the use of oral contraceptives, hormone replacement therapy, or gonadotropin-releasing hormone agonists/antagonists.
  2. Premenopausal or perimenopausal (perimenopause defined as age ≥50 to <60 years, with amenorrhea <12 months or FSH and/or E2 not within the postmenopausal range): must initiate ovarian function suppression with a luteinizing hormone-releasing hormone agonist (e.g., goserelin or leuprolide) ≥2 weeks prior to Day 1 of Cycle 1 and continue throughout the study.
* A tumor tissue test report confirming the presence of a PIK3CA mutation must be available.
* Provision of fresh tumor tissue (preferred) or archived tumor tissue collected within 2 years.
* At least one measurable lesion as assessed by RECIST v1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Estimated life expectancy ≥3 months.
* Adequate hematologic and organ function within 7 days prior to the first dose of GenSci145,as Hematology,Hepatic Function,Renal Function,Glucose Metabolism,Coagulation.
* Women of childbearing potential (WOCBP) must voluntarily agree to use adequate contraception from the time of signing the ICF until at least 60 days after the last dose of GenSci145 (or up to 2 years if in combination with fulvestrant, in accordance with local prescribing information), and must have a negative serum human chorionic gonadotropin (hCG) test within 7 days prior to the first dose of GenSci145.
* Male participants with reproductive potential must voluntarily agree to use adequate contraception from the time of signing the ICF until at least 98 days after the last dose of GenSci145 (or up to 2 years if in combination with fulvestrant, in accordance with local prescribing information).

Exclusion Criteria:

* History of any active malignancy within ≤2 years prior to the first dose of GenSci145, except for the malignancy under investigation in this study and any curatively treated locally recurrent malignancies
* Presence of symptomatic, untreated, or progressing CNS metastases. Participants with previously treated CNS metastases (e.g., by surgery or radiotherapy) are eligible only if all of the following conditions are met:

  1. Disease stable for at least 3 months, with no evidence of progression on imaging within 4 weeks prior to first dose of study treatment, all neurologic symptoms recovered to baseline, and no evidence of new or enlarging brain metastases.
  2. At least 4 weeks have elapsed since completion of CNS-directed radiotherapy, surgery, or corticosteroid therapy prior to the first dose of study treatment.
* History of leptomeningeal metastases, spinal cord compression, or leptomeningeal disease.
* History of acute pancreatitis (within 1 year) or chronic pancreatitis, or radiologic evidence of pancreatic metastases.
* History of stroke, transient ischemic attack, or other clinically significant cerebrovascular events within 6 months prior to the first dose of GenSci145.
* Active infection requiring intravenous antibiotics, or other uncontrolled intercurrent illness requiring hospitalization. Minor infections such as periodontal infection or urinary tract infection manageable with short-course oral antibiotics are permitted.
* Confirmed diagnosis of uncontrolled diabetes mellitus, defined as HbA1c ≥8% and/or fasting plasma glucose ≥140 mg/dL (7.7 mmol/L).
* Uncontrolled hypertension, defined as blood pressure ≥150/90 mmHg despite optimal medical management.
* Clinically significant cardiovascular disease, including but not limited to:

  1. Myocardial infarction or unstable angina within 6 months prior to the first dose of GenSci145.
  2. New York Heart Association (NYHA) Class III or higher within 4 weeks prior to the first dose.
  3. Left ventricular ejection fraction (LVEF) <50%, assessed by echocardiogram within 4 weeks prior to the first dose.
  4. Based on three consecutive resting ECGs collected during the screening, the average QT interval corrected by Fridericia's formula (QTcF) is >450 ms for males and >470 ms for females.

     Any condition associated with increased risk of torsades de pointes (e.g., persistent hypokalemia despite standard treatment, family
  5. history of long QT syndrome).
  6. Any clinically significant cardiac rhythm, conduction, or resting ECG abnormality (e.g., complete left bundle branch block, second- or third-degree atrioventricular block).
* Interstitial lung disease, drug-induced pneumonitis, radiation pneumonitis requiring corticosteroid treatment, or other severe pulmonary diseases affecting lung function.
* Gastrointestinal disorders that, in the opinion of the investigator, may interfere with the absorption of oral GenSci145, such as peptic ulcer disease, uncontrolled nausea or vomiting, malabsorption syndrome, history of small bowel resection, or active inflammatory bowel disease (e.g., Crohn's disease or ulcerative colitis).
* Uncontrolled serosal effusion, including pleural effusion, ascites, or pericardial effusion (participants with effusions that are controlled and stable for ≥2 weeks after treatment may be eligible).
* Prior treatment with PI3K, mTOR, or AKT inhibitors.
* Prior treatment with fulvestrant (except in Phase 1a and Part 4 Cohort 4).
* Receipt of a live attenuated vaccine within 4 weeks prior to the first dose of GenSci145.
* Prior anticancer therapies before the first dose of GenSci145 as follows:

  1. Herbal medicines or traditional Chinese medicines with antitumor activity within 2 weeks
  2. Endocrine therapy with antitumor indications within 2 weeks or 5 half-lives (whichever is shorter).
  3. Radiotherapy within 4 weeks.
  4. Chemotherapy within 4 weeks (≥6 weeks for nitrosoureas or mitomycin; oral fluoropyrimidines allowed within 14 days or 5 half-lives, whichever is longer).
  5. Small molecule targeted agents, biologics, or immunotherapy within 4 weeks or 5 half-lives (whichever is shorter).
* Major surgery within 4 weeks prior to the first dose of GenSci145, or currently recovering from surgery, or planned major surgery during the study.
* Use of strong inducers or inhibitors of cytochrome P450 3A4 (CYP3A4), or drugs known to prolong the QT/QTc interval, within 5 half-lives or 14 days before the first administration of GenSci145.

Current or recent systemic corticosteroid therapy, or not fully recovered from adverse reactions of prior systemic corticosteroid use (local administration permitted, e.g., topical for rash, inhalation for COPD, 19.ophthalmic use, or intra-articular injection).

* History of organ transplantation or allogeneic stem cell transplantation.
* Inability to swallow oral medications (e.g., tablets or capsules) without chewing, breaking, crushing, opening, or otherwise altering the product form.

  22.Positive test results for hepatitis B virus (HBsAg positive; participants must also undergo HBV DNA testing, and levels above the assay ULN will result in exclusion), hepatitis C virus (HCV Ab positive; participants must also undergo HCV RNA testing, and levels above the assay ULN will result in exclusion), or human immunodeficiency virus (HIV Ab positive).
* Persistent toxicities from prior anticancer therapy of CTCAE v6.0 Grade ≥2 (except for alopecia and ≤Grade 2 peripheral sensory neuropathy, or other ≤Grade 2 adverse events deemed not to pose a safety risk by the investigator).
* Known severe hypersensitivity to GenSci145 and/or any of its excipients; for participants in combination cohorts, known hypersensitivity to fulvestrant or to palbociclib (applicable to Part 3 triplet and Part 4 Cohort 3).
* Pregnant or breastfeeding women, or women planning to breastfeed during the study or within 60 days after the last dose of GenSci145 (or up to 2 years if in combination with fulvestrant, in accordance with local prescribing information).
* Participation in another clinical study within 4 weeks prior to the first dose (except for observational, non-interventional studies or participants in the follow-up phase of an interventional trial).

Any other condition that, in the opinion of the investigator, would make the participant unsuitable for study participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2026-03-14 (Estimated); Primary Completion 2028-11-08 (Estimated); Study Completion 2029-02-21 (Estimated)

PRIMARY OUTCOMES:
Phase Ia :Incidence and severity of treatment-emergent adverse events (TEAEs) | Collect the adverse events (AES) that occurred in the subjects from the signing of the ICF to 30 days after the last administration of the investigational drug or the initiation of a new anti-tumor treatment (whichever occurs first).
Part1:Dose limiting toxicities(DLTs) | At the end of Cycle 1 (each cycle is 28 days).

SECONDARY OUTCOMES:
To determine the maximum tolerated dose (MTD) (if applicable) and recommended dose for expansion (RDE) of GenSci145. | Approximately form time of first dose of GenSci145 up to 12 months.
Peak concentration (Cmax) of GenSci145 | Approximately 12 months.
Peak time (Tmax) of GenSci145 | Approximately 12 months.
The area under the drug-time curve from time 0 to the last measurable concentration time point (AUC0-last) of GenSci145 | Approximately 12 months.
Half-life (t1/2) of GenSci145 | Approximately 12 months.
Apparent clearance rate (CL/F) of GenSci145 | Approximately 12 months.
The apparent distribution volume (Vd/F) and the area under the drug-time curve from time 0 to infinity (AUC0-inf) of GenSci145. | Approximately 12 months.
ORR,the best overall response (BOR) is achieved at complete response (CR) or partial response (PR) Proportion of subjects. | Approximately 12 months.

OTHER OUTCOMES:
DOR,from the first assessment of CR or PR to the first assessment of disease progression (PD) or death The duration of (whichever occurs first). | Approximately 12 months.
DCR,the proportion of subjects whose BOR reached CR, PR or disease stability (SD). | Approximately 12 months.
CBR,the proportion of subjects whose BOR reached CR, PR or SD (duration ≥6 months). | Approximately 12 months.
TTR,the time from the first treatment to the first assessment of CR or PR. | Approximately 12 months.
:PFS ,the date from the first treatment to the first occurrence of PD or death (whichever occurs first). | Approximately 12 months.
OS ,the date from the first treatment to death for any reason. | Approximately 12 months.

CONTACTS AND LOCATIONS:
Locations (1):
- The Cancer Hospital of the Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China